CLINICAL TRIAL: NCT01435811
Title: Dose Range Evaluation of Norovirus Challenge Pool (GII.4, CIN-1)
Acronym: CIN-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: LigoCyte Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: CIN-002
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Norovirus Infections
Keywords: Norovirus
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norovirus challenge pool (GII.4, CIN-1) (Experimental)
  Interventions: Biological: Norovirus challenge pool (GII.4, CIN-1)
- Sterile water (Placebo Comparator)
  Interventions: Biological: Norovirus challenge pool (GII.4, CIN-1)

INTERVENTIONS:
Biological: Norovirus challenge pool (GII.4, CIN-1) — Norovirus challenge pool (GII.4, CIN-1)

SUMMARY:
The purpose of this study is to determine a suitable dose of the human norovirus GII.4 challenge pool(CIN-1;031693) that induces illness in approximately 50% of susceptible subjects that would be useful for evaluation of vaccines and antivirals.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between the ages of 18 and 49 years
2. Willing and able to provide written informed consent
3. Able to comply with all study procedures
4. Have a serum antibody titer of < 1:1600 to the GII.4 challenge strain of Norovirus as measured by ELISA
5. Female subjects of childbearing potential must have negative urine pregnancy tests, at screen and prior to challenge
6. Female subjects must be of non-childbearing potential, or if of childbearing potential (as determined by investigator) must be practicing abstinence or using an effective licensed method of birth control (e.g. oral contraception; diaphragm or condom in combination with contraceptive jelly, cream, or foam; intrauterine contraceptive device, or hormonal devices/injections (for example, NORPLANT® or DEPO-PROVERA®) from screening through one month after completing inpatient stay.
7. Have normal screening laboratories for SGPT (ALT), creatinine, sodium, potassium, total white blood cell count (WBC), hemoglobin, neutrophils, lymphocytes, platelets, urine protein, urine glucose and urine RBCs (see table below) as well as negative stool culture for known bacterial pathogens and stool evaluation for parasites.
8. For challenged subjects: Be secretor positive for HBGA binding by assay of their saliva. For placebo recipients: Be secretor negative for HBGA binding by assay of their saliva.
9. Score at least 70% on a test of understanding of this research study.

Exclusion Criteria:

* Expected to be noncompliant with study procedures or planning to move within the anticipated total duration of the study (180 days after challenge)
* Pregnant or breastfeeding
* HIV positive (by history or screening antibody test)
* Hepatitis B positive (by history or a positive hepatitis B surface antigen)
* Hepatitis C positive (by history or a positive antibody to hepatitis C virus)
* Norovirus GII.4 serum antibody screening titer of > 1:1600
* Clinically significant findings on history or physical examination
* Temperature >38.00C, resting heart rate >100/beats per minute or <55/beats per minute, systolic blood pressure >140, diastolic blood pressure >90, systolic blood pressure <90, respiratory rate >16/min. If heart rate <55 beats per minute and investigator determines that this is not clinically significant and heart rate increases > 55 beats per minute on moderate exercise (two flights of stairs), subject will not be excluded. Vital signs may be repeated at screening.
* Clinically significant history of diseases or treatments that may affect the immune system's function such as a past history of cancer, receipt of chemotherapy or radiation therapy, or autoimmune diseases (exception; a history of basal cell or squamous cell carcinoma in remission without treatment for more than 5 years prior to study entry)
* Receipt of systemic corticosteroids for greater than 7 days within the past six months
* Clinically abnormal screening electrocardiogram (ECG) defined as pathologic Q waves and significant ST-T wave changes: criteria for left ventricular hypertrophy; and any non-sinus rhythm excluding isolated premature atrial contractions
* Clinically significant respiratory disease, endocrine disease, liver disease, renal disease, or neurological disease
* History of malabsorption or maldigestion disorder (e.g. celiac sprue), major gastrointestinal (GI) surgery, or any other chronic GI disorders that would interfere with the study
* Clinically significant abnormalities of the health screening laboratory work
* Use of antibiotics within 7 days prior to entry into the inpatient facility (Day -1)
* Any chronic medical illness requiring a new prescription medication or hospitalization during the screening period.
* Temperature ≥38.0°C or self-reported diarrhea or vomiting during the 7 days prior to challenge administration (Day 0)
* History of treatment within the past year for an eating disorder
* Self-reported history of alcohol or drug abuse within past 3 years
* Receipt of any vaccine, licensed or investigational, or any investigational product within 30 days of challenge administration or plan to receive any vaccine or investigational product through up to one month after leaving the inpatient facility
* Use of any H2 receptor antagonists (e.g., Tagamet, Zantac, and Pepcid), proton pump inhibitors (e.g., Prilosec, OTC, Protonix, and Prevacid), or prescription acid suppression medication or over-the-counter (OTC) antacids within 72 hours of investigational product administration (Day 0)
* Use of prescription and OTC medications containing acetaminophen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs within 48 hours prior to investigational product administration (Day 0)
* Regular use of laxatives or anti-motility agents
* Receipt of blood or blood products within the past six months
* Subjects who are unwilling or unable to cease smoking for the duration of the inpatient stay
* Any other condition, such as a medical, psychiatric, or social condition or occupational responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to the subject's participation in the study or assessment of the investigational product
* Plan to be living in a confined environment (e.g. ship, camp, or dormitory) within 3 weeks after receiving the challenge strain
* Commercial food handlers, day care workers, or health care workers involved in direct patient contact
* Provide child day care services either in a home or in a nonresidential facility
* Provide direct care to individuals over 65 years of age
* Subjects with young children (<2 years) at home or with household contacts who are:

  * Immunocompromised
  * Pregnant, or
  * Breast feeding

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Dose range evaluation of Norovirus challenge pool (GII.4, CIN-1) | 6 months
  To determine a suitable dose of the human norovirus GII.4 challenge pool (CIN-1;031693) that induces illness in approximately 50% of susceptible subjects that would be useful for evaluation of vaccines and antivirals.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States